CLINICAL TRIAL: NCT06632470
Title: Clinical Utility and Safety of Human Umbilical Cord Mesenchymal Stem Cell Secretome in Moderate Neurocognitive Impairment (Dementia)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baermed (Other)
Collaborators: Tarumanagara University (Other); panti werda hana (Unknown); LPPT TARUMANAGARA (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 018-UTHREC/UNTAR/VIII/2024
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Dementia; Moderate Dementia
Keywords: dementia; moderate dementia; neurocognitive impairment; secretome; HUCSMC; stem cells
MeSH Terms: conditions — Dementia | interventions — Secretome; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Secretome injection (Experimental): patient will receive secretome injection every two weeks for four months
  Interventions: Drug: Secretome injection
- Vitamin B12 (Placebo Comparator): patient will receive 1 ampule of vitamin b12 every two weeks for 4 months
  Interventions: Drug: Vitamin B12 Injection

INTERVENTIONS:
Drug: Secretome injection — Patient will receive 3 ml of secretome intramuscular injection every two weeks for four months
  Other Names: secretome; hucmsc
  Arms: Secretome injection
Drug: Vitamin B12 Injection — Patient will receive 1 ampule of vitamin b 12 intramuscular injection as a placebo drug every two weeks for four months
  Arms: Vitamin B12

SUMMARY:
The goal of this clinical trial if to learn if Human Umbilical Cord Mesenchymal Stem Cell (HUCMSC) derived secretome injection is safe and effective in patient with moderate dementia. The main questions it aims to answer are:

1. Is HUCMSC derived secretome safe to be use as a therapy in patients with moderate dementia?
2. How does HUCMSC derived secretome affect pro inflammatory and anti inflammatory cytokine (IL-6 and TNF alfa) in patient with moderate dementia?
3. What is the relationship between HUCMSC derived secretome therapy with mini mental state examination? Researchers will compare the intervention group (patients who are injected with HUCMSC derived secretome) and control group (patients who are only monitored)

Participants will

* Be injected with HUCMSC derived secretome or Vitamin B12 every two weeks for 4 months
* Follow up visit to review treatment progress on 3rd months (2 weeks post treatment), 7th months (3 months post treatment) and participants will do several blood test and mental examination

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years old
2. Patient diagnosed with dementia confirmed by psychiatrist or neurologist based on DSM-4 or ICD 10
3. Patient with Mini-Mental State Examination (MMSE) between 10 to 20 indicating moderate cognitive impairment
4. Patient is in stable condition without life threatening disease or uncontrolled medical condition
5. Patient undergoing stable dose treatment for other medical condition at least 4 months before the trial
6. Patient with care giver or supporting family who can assist patient with research protocol

Exclusion Criteria:

1. Patient has dementia due to other medical condition such as severe head trauma, brain infection or history of drug abuse
2. Patient with uncontrolled medical condition such as severe cardiovascular disease, chronic lung disease, cancer, or systemic infection
3. Patient with severe psychiatry disorder such as schizophrenia and bipolar disorder
4. Patient is receiving experimental drugs or participates in experimental studies for the last 30 days before the trial
5. Patient who has allergy or hypersensitivity reaction towards secretome
6. Patient with medical complications or surgery complications that require immediate interventions or other life threatening complications
7. Patient is unable to provide written informed consent and not capable to understand and comply to research protocol
8. Patient is unwilling and not capable to follow research protocol including follow up evaluations and blood sampling according to schedule

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of moderate dementia patients with normal range of blood parameters assessed by hemoglobin level, hematocrit level, leukocyte level, thrombocyte level, HbA1c level, kidney function and liver function | From enrollment to 3 months after treatment
  The blood parameters such as hemoglobin, hematocrit, leukocyte, thrombocyte, HbA1c, kidney function and liver function normal range is measured according to international standard
Number of participants with improved Mini mental status examination, mini cog and AD8 | from enrollment to 3 months after treatment
  Participants achieved a response if they have improvement of MMSE score, mini cog score and AD8 score
Number of participants with improved Glial Fibrillary Acid Protein (GFAP) levels | from enrollment to 3 months after treatment
  Participants achieved a response if there is a decrease in GFAP levels

CONTACTS AND LOCATIONS:
Overall Officials: Noer Saelan Dr. dr. Noer Saelan Tadjudin Sp.KJ, Principal Investigator — Tarumanagara University
Locations (1):
- Panti Werda Hana, Tangeran Selatan, Banten, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Case Report Form (all collected IPD)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication with no end date

REFERENCES:
- [Background] Chiu EC, Chien TH, Lee YC. Measurement Equivalence between the Original and Estimated Mini-Mental State Examination in People with Dementia. Int J Environ Res Public Health. 2021 Jul 17;18(14):7616. doi: 10.3390/ijerph18147616. PMID 34300067
- [Background] Myrberg K, Hyden LC, Samuelsson C. The mini-mental state examination (MMSE) from a language perspective: an analysis of test interaction. Clin Linguist Phon. 2020 Jul 2;34(7):652-670. doi: 10.1080/02699206.2019.1687757. Epub 2019 Nov 18. PMID 31739693
- [Background] Arevalo-Rodriguez I, Smailagic N, Roque I Figuls M, Ciapponi A, Sanchez-Perez E, Giannakou A, Pedraza OL, Bonfill Cosp X, Cullum S. Mini-Mental State Examination (MMSE) for the detection of Alzheimer's disease and other dementias in people with mild cognitive impairment (MCI). Cochrane Database Syst Rev. 2015 Mar 5;2015(3):CD010783. doi: 10.1002/14651858.CD010783.pub2. PMID 25740785
- [Background] Thanaskody K, Jusop AS, Tye GJ, Wan Kamarul Zaman WS, Dass SA, Nordin F. MSCs vs. iPSCs: Potential in therapeutic applications. Front Cell Dev Biol. 2022 Nov 2;10:1005926. doi: 10.3389/fcell.2022.1005926. eCollection 2022. PMID 36407112
- [Background] Lee C, Kim M, Han J, Yoon M, Jung Y. Mesenchymal Stem Cells Influence Activation of Hepatic Stellate Cells, and Constitute a Promising Therapy for Liver Fibrosis. Biomedicines. 2021 Nov 2;9(11):1598. doi: 10.3390/biomedicines9111598. PMID 34829827
- [Background] Teixeira FG, Panchalingam KM, Assuncao-Silva R, Serra SC, Mendes-Pinheiro B, Patricio P, Jung S, Anjo SI, Manadas B, Pinto L, Sousa N, Behie LA, Salgado AJ. Modulation of the Mesenchymal Stem Cell Secretome Using Computer-Controlled Bioreactors: Impact on Neuronal Cell Proliferation, Survival and Differentiation. Sci Rep. 2016 Jun 15;6:27791. doi: 10.1038/srep27791. PMID 27301770
- [Background] Willis CM, Nicaise AM, Hamel R, Pappa V, Peruzzotti-Jametti L, Pluchino S. Harnessing the Neural Stem Cell Secretome for Regenerative Neuroimmunology. Front Cell Neurosci. 2020 Nov 5;14:590960. doi: 10.3389/fncel.2020.590960. eCollection 2020. PMID 33250716
- [Background] Park JH, Jung SJ, Lee LJ, Rhu J, Bae SH. Impact of nonpharmacological interventions on cognitive impairment in women with breast cancer: A systematic review and meta-analysis. Asia Pac J Oncol Nurs. 2023 Mar 1;10(4):100212. doi: 10.1016/j.apjon.2023.100212. eCollection 2023 Apr. PMID 37095894
- [Background] Treanor CJ, McMenamin UC, O'Neill RF, Cardwell CR, Clarke MJ, Cantwell M, Donnelly M. Non-pharmacological interventions for cognitive impairment due to systemic cancer treatment. Cochrane Database Syst Rev. 2016 Aug 16;2016(8):CD011325. doi: 10.1002/14651858.CD011325.pub2. PMID 27529826
- [Background] Hafiz R, Alajlani L, Ali A, Algarni GA, Aljurfi H, Alammar OAM, Ashqan MY, Alkhashan A. The Latest Advances in the Diagnosis and Treatment of Dementia. Cureus. 2023 Dec 14;15(12):e50522. doi: 10.7759/cureus.50522. eCollection 2023 Dec. PMID 38222245
- [Background] Salomone S, Caraci F, Leggio GM, Fedotova J, Drago F. New pharmacological strategies for treatment of Alzheimer's disease: focus on disease modifying drugs. Br J Clin Pharmacol. 2012 Apr;73(4):504-17. doi: 10.1111/j.1365-2125.2011.04134.x. PMID 22035455
- [Background] Pierre G. Neurodegenerative disorders and metabolic disease. Arch Dis Child. 2013 Aug;98(8):618-24. doi: 10.1136/archdischild-2012-302840. Epub 2013 May 22. PMID 23698595
- [Background] Zriek F, Di Battista JA, Alaaeddine N. Mesenchymal Stromal Cell Secretome: Immunomodulation, Tissue Repair and Effects on Neurodegenerative Conditions. Curr Stem Cell Res Ther. 2021;16(6):656-669. doi: 10.2174/1574888X16666210202145639. PMID 33530914
- [Background] Guo J, Huang X, Dou L, Yan M, Shen T, Tang W, Li J. Aging and aging-related diseases: from molecular mechanisms to interventions and treatments. Signal Transduct Target Ther. 2022 Dec 16;7(1):391. doi: 10.1038/s41392-022-01251-0. PMID 36522308
- [Background] Morrone A, Donini LM, Scardella P, Piombo L, Pinto A, Giusti AM, Neri B, Hagedorn T, Proietti AR, Cataldi S, Cucinotta D, Di Bella G, Barbagallo M, Cannella C; Gruppo di Lavoro MEG. [Malnutrition in the elderly: clinical features, psychological and social determinants. Preliminary results]. Ann Ig. 2011 Mar-Apr;23(2):161-72. Italian. PMID 21770232
- [Background] Bhatia MS, Srivastava S, Moond V. Prevalence of cognitive dysfunction, psychological morbidity and abuse in the community-based elderly population in India. Gen Psychiatr. 2020 Aug 16;33(5):e100207. doi: 10.1136/gpsych-2020-100207. eCollection 2020. PMID 32875272
- [Background] Ezkurdia A, Ramirez MJ, Solas M. Metabolic Syndrome as a Risk Factor for Alzheimer's Disease: A Focus on Insulin Resistance. Int J Mol Sci. 2023 Feb 22;24(5):4354. doi: 10.3390/ijms24054354. PMID 36901787
- [Background] Emmady PD, Schoo C, Tadi P. Major Neurocognitive Disorder (Dementia). 2022 Nov 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557444/ PMID 32491376
- [Background] Rasmussen KL, Frikke-Schmidt R. The current state of apolipoprotein E in dyslipidemia. Curr Opin Lipidol. 2024 Apr 1;35(2):78-84. doi: 10.1097/MOL.0000000000000915. Epub 2023 Dec 6. PMID 38054895
- [Background] Shen C, Liu C, Qiu A. Metabolism-related brain morphology accelerates aging and predicts neurodegenerative diseases and stroke: a UK Biobank study. Transl Psychiatry. 2023 Jun 29;13(1):233. doi: 10.1038/s41398-023-02515-1. PMID 37385998
- See also: Related Info — https://journals.eco-vector.com/RFD/article/view/70198/en_US
- See also: Related Info — https://openalex.org/works/W4283263957
- See also: Related Info — https://link.springer.com/chapter/10.1007/978-3-319-44775-9_3